CLINICAL TRIAL: NCT00064532
Title: Serum Sex Hormone Levels and Subclinical Atherosclerosis - Ancillary to MESA
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Kiang Liu, Professor in Preventive Medicine and Geriatrics and Internal Medicine, Northwestern University
Other Study IDs: 1226; R01HL074338 (NIH)
Record Dates: First submitted 2003-07-08; First posted 2003-07-10 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2013-11

CONDITIONS: Cardiovascular Diseases; Atherosclerosis; Coronary Arteriosclerosis; Coronary Disease; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Coronary Artery Disease; Coronary Disease; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
To assess the associations of serum sex hormones with the presence and progression of subclinical atherosclerosis.

DETAILED DESCRIPTION:
BACKGROUND:

Throughout their lifetime, men are at higher risk of coronary heart disease (CHD) than women, however, after menopause this difference is attenuated. This observation suggests that endogenous sex hormones could be associated with CHD risk. There is some evidence indicating that the effect of sex hormones on CHD risk could be mediated, in part, by alterations in lipid levels or other CHD risk factors. However, other evidence supports an independent relationship of circulating hormone levels with CHD risk.

DESIGN NARRATIVE:

The study, which is ancillary to MESA, will examine the associations of serum sex hormone concentrations with the presence and progression of subclinical atherosclerosis in 3,259 male and 2,802 postmenopausal female participants of the Multi-Ethnic Study of Atherosclerosis (MESA). Subclinical atherosclerosis will be identified using both coronary artery calcium (CAC) and carotid intimal-medial wall thickness (IMT). Progression will be identified by the change in CAC over 3.5 years. Circulating concentrations of total (and free) testosterone (T), dehydroepiandrosterone (DHEA), 17 beta-estradiol (E2), and sex hormone binding globulin (SHBG) in stored serum samples collected at the MESA baseline exam will be assessed. Laboratory results will be merged with existing demographic, anthropometric, lifestyle, CHD risk factor, and subclinical disease data collected in MESA. Cross-sectional and prospective methods of statistical analysis will be used to assess the proposed associations. MESA is particularly well suited for disentangling the effects of hormonal factors and CHD risk factors on subclinical atherosclerosis because of the availability of high-quality data, serum samples, and CAC and IMT measurements in a large multi-ethnic population of men and women.

ELIGIBILITY:
Exclusion Criteria:

* Age younger than 45 or older than 84 years
* Physician-diagnosed heart attack
* Physician-diagnosed angina or taking nitroglycerin
* Physician-diagnosed stroke or TIA
* Physician-diagnosed heart failure
* Current atrial fibrillation
* Having undergone procedures related to cardiovascular disease (CABG, angioplasty, valve replacement, pacemaker or defibrillator implantation, any surgery on the heart or arteries)
* Active treatment for cancer
* Pregnancy
* Any serious medical condition which would prevent long-term participation
* Weight >300 pounds
* Cognitive inability as judged by the interviewer
* Living in a nursing home or on the waiting list for a nursing home
* Plans to leave the community within five years
* Language barrier (speaks other than English, Spanish, Cantonese or Mandarin)
* Chest CT scan in the past year

Ages: 45 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample of African-American, Chinese-American, Caucasian, and Hispanic residents drawn from six regions in the United States: Baltimore City and Baltimore County, Maryland; Chicago, Illinois; Forsyth County, North Carolina; Los Angeles County, California; New York, New York; and St. Paul, Minnesota.
Sampling Method: Non-Probability Sample
Enrollment: 6173 (Actual)
Dates: Start 2003-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Coronary artery calcium | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Susan Gapstur, Principal Investigator — Northwestern University